CLINICAL TRIAL: NCT03454100
Title: Community Resilience to Acute Malnutrition
Acronym: CRAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Concern Worldwide (Unknown); Department for International Development, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A06/B14
Record Dates: First submitted 2018-02-09; First posted 2018-03-05 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-02

CONDITIONS: Malnutrition, Child
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: Panel cluster randomized intervention trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multi-sectoral package of activities (Experimental): Villages in the experimental arm received the full multi-sectoral package of village level activities, including having a well dug, a shared latrine installed, training on handwashing and hygiene across the water chain, training on conservation agriculture techniques, care groups for pregnant and breastfeeding mothers, and training on market gardens.
  Interventions: Behavioral: multisectoral package of activities
- Control (No Intervention): Villages in the control arm did not receive teh multi-sectoral package of village level activities.

INTERVENTIONS:
Behavioral: multisectoral package of activities — A multi-sectoral package of village level activities, including having a well dug, a shared latrine installed, training on handwashing and hygiene across the water chain, training on conservation agriculture techniques, care groups for pregnant and breastfeeding mothers, and training on market gardens.
  Arms: multi-sectoral package of activities

SUMMARY:
The study evaluates the impact of a multi-sectoral intervention (water, sanitation, and hygiene; training on climate smart activities; care groups for mothers; market gardens) on the prevalence of acute malnutrition as the primary outcome using a randomized intervention trial between 2012-2017 with four points of data collection (2012, 2014, 2015, and 2017).

DETAILED DESCRIPTION:
Concern Worldwide has developed a model of intervention called Community Resilience to Acute Malnutrition (CRAM). This model is based on the need for (a) the introduction of longer-term programming to build community resilience to shocks, while recognising that there may be a need for humanitarian intervention, and (b) a multi-sectoral package of activities given experience in programming from other settings. The goal of the study is to rigorously test the impact of the model and associated activities on community resilience to shocks in the Goz Beida area of Chad. Where community resilience is proxied by the primary outcome variable: acute malnutrition.

In order to answer this question, 69 villages had been randomized to either receive the full multi-sectoral program or not. In each village, approximately 20 households were surveyed (randomly selected from a household list from a previous emergency distribution) for a total of 1420 households. Those households were then surveyed in November/December 2012 (prior to the intervention), and again a the same time period in 2014, 2015, and 2017.

Data was collected on household demographics, livelihoods, child health, and nutrition, including child (6-59 months) anthropometry.

ELIGIBILITY:
Inclusion Criteria:

* child is from household with B, C, or D wealth ranking (wealth ranking is from A-D with A being the highest wealth and D being the lowest wealth)
* child is between the ages of 6-59 months
* child is present in the selected household at the time of the survey

Exclusion Criteria:

* child has a skin disorder
* too ill to be measured on height board or weight scale

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1420 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Acute Malnutrition | 5 years
  prevalence of wasting (weight for age z-score<-2)

SECONDARY OUTCOMES:
Chronic Malnutrition | 5 years
  prevalence of stunting (height for age z-score<-2)
height for age | 5 years
  height for age z-score
child morbidity | 5 years
  Child ill in the past two weeks
weight for height | 5 years
  weight for height z-score

CONTACTS AND LOCATIONS:
Overall Officials: Helen Young, DR, Principal Investigator — Tufts University
Locations (1):
- Concern Worldwide Office, Goz Beida, Sila Region, Chad

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marshak A, Young H, Bontrager EN, Boyd EM. The Relationship Between Acute Malnutrition, Hygiene Practices, Water and Livestock, and Their Program Implications in Eastern Chad. Food Nutr Bull. 2017 Mar;38(1):115-127. doi: 10.1177/0379572116681682. Epub 2016 Dec 8. PMID 27932595